CLINICAL TRIAL: NCT04964999
Title: Microgravity Research Analogue (MRA): Understanding the Health Impact of Inactivity for the Benefit of Older Adults and Astronauts Initiative
Brief Title: Understanding the Negative Effects of Bed Rest and Using Exercise as Countermeasure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Space Agency (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Jose Morais, Professor and Director, Division of Geriatric Medicine, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MP-37-2021-7170
Record Dates: First submitted 2021-05-06; First posted 2021-07-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Aging
Keywords: Bed rest; Exercise; Aging
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled study - Participants will be randomly allocated to the exercise or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will perform aerobic and strength exercises for 2 weeks.
  Interventions: Other: Exercise
- No exercise (No Intervention): Participants will not perform any exercises.

INTERVENTIONS:
Other: Exercise — Participants will undergo an exercise program during the 2-week bed rest period.
  Arms: Exercise

SUMMARY:
Physical activity appears to be an important lifestyle habit to achieve healthy aging by promoting autonomy and quality of life. Interestingly, the dramatic changes that the human body undergoes due to bedrest for illnesses and hospitalization are similar to those seen over decades of normal aging. Bedrest in otherwise healthy older individuals can lead to a reduction of muscle size and strength, changes in bone strength and function of the heart and blood vessels. Bedrest can also lead to changes in keeping proper balance as well as changes in processing and understanding information. All of these factors negatively affect activities of daily living leading to physical function impairment and development of frailty, a clinical condition associated with an increased risk for disease and death.

The purpose of this study is to investigate whether exercise can counteract the negative effects of 2-week head tilt down bed rest on muscle function and metabolism, postural control, bone structure, orthostatic tolerance and cognitive function in adults.

For this study the investigators will recruit 24 healthy men and women between 55 - 65 years of age. All subjects will spend a total of 26 days (5 days of adaption period, 14 days of bed rest with 6 degrees of downward inclination, and 7 days of recovery period) at the McGill University Health Centre (MUHC). During this study, 12 subjects will randomly undergo an exercise intervention as countermeasure during the 14 days of bed rest period and 12 will serve as control.

Each subjects participation in this study will involve 1 telephone call (pre-screening) and 4 visits at the MUHC: 1 screening visit (Visit 1) followed by a 26-day long visit (Visit 2) and 2 follow-up visits (Visit 3 and Visit 4). During Visits 2 - 4 various measurements will be performed to assess sensorimotor control, muscle function and metabolism, bone structure, cardiovascular function, cognitive performance and function, and specimen collection (blood, urine, saliva, feces and muscle tissue).

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 20 and a maximum of 24 non-smoking participants in the age group of 55 to 65 years old, half male and half female.
* Female participants must be menopausal (no menses for at least 1 year (or documented ovariectomy) and a serum FSH above 30 IU/L).
* Height between 158 to 190 cm with a body mass index between 20 to 30 kg/m2.
* Physically and mentally healthy subjects that will have successfully passed the psychological and medical screening appropriate for the age group.
* Participation in at least 2.5 hours of exercise at a moderate to vigorous-intensity aerobic activity per week.
* Willing to be assigned randomly either to the exercise or the control group.

Exclusion Criteria:

* Participants must be dementia-free, drug- or alcohol-addiction free, with no history of heart attacks, no thrombosis risk, no severe allergies, no hypocalcaemia, no uric acidemia, no orthostatic intolerance, no vestibular disorders, no considerable musculoskeletal issues, no chronic back pain, no head trauma, no seizures, no ulcers, no renal stones, no gastro-esophageal reflux disease or renal function disorder, no hiatus hernia, no migraines, and no mental illness.
* Electrocardiogram abnormalities
* Anemia
* Low bone mineral density
* Medication requirements that may interfere with the interpretation of the results
* Recent substandard nutritional status
* Claustrophobia
* Special dietary requests (e.g. vegetarian, vegan or some other diet)
* Sedentary people and people that are addicted to exercise
* Metallic implants (pacemakers, ICDs, CRT devices, infusion pumps, cerebral artery aneurysm clips, dental implants, tissue expander etc.), osteosynthesis material
* Given blood in the past 3 months before the onset of the experiment
* Smoked (tobacco and/or marijuana (THC)) within 6 months prior to the start of the study
* Abused drugs, medicine or alcohol within up to 30 days prior to the start of the study
* Participated in another study within 2 months before study onset

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Changes in cognition status of participants with head down bed rest (HDBR) with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  NIH Toolbox Cognition Battery (computerized)
Changes in cognition status of participants with head down bed rest (HDBR) with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  CLSA cognition questionnaire
Changes in emotional status of participants with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Positive and Negative Affect Scale
  - For both scales scores can range from 10-50, with higher scores representing higher levels of positive or negative affect.
Changes in emotional status of participants with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  General Health Questionnaire (GHQ-28).
  * Using Likert 4-point scale with the min score being 0 and max score being 84.
  * Higher scores indicate a higher level of distress.
Changes in brain structure with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Assessment of brain anatomy using a MRI.
Changes in brain function with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Measurement of neuronal, cerebrovascular, and connectivity integrity with functional MRI.
Changes in muscle muscle mass with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Body MRI
Changes in muscle fat infiltration with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Body MRI
Changes in adiposity with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Body MRI
Changes in ventricular volume of the heart with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using a heart MRI left and right ventricular volumes will be assessed.
Changes in ventricular mass with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using a heart MRI left and right ventricular mass will be assessed.
Changes in bone structure with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  High resolution peripheral quantitative computed tomography (HR-pQCT)
Changes in muscle strength with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Quantitative Muscle Dynamometry (Biodex)
Changes in muscle strength with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Vertical jump
Changes in muscle-pump baroreflex with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Supine-to-stand test
Changes in balance control with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Postural equilibrium control test
Changes in orthostatic tolerance with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Tilt test
Cardiac and vascular changes with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using high frame rate ultrasound (HiFRUS) arterial wall shear stress will be assessed.
Cardiac and vascular changes with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using high frame rate ultrasound (HiFRUS) arterial wall stiffness will be assessed.
Cardiac and vascular changes with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using high frame rate ultrasound (HiFRUS) cardiac mass will be assessed.
Cardiac and vascular changes with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using high frame rate ultrasound (HiFRUS) patterns of blood flow will be assessed.
Changes in Fractional Synthesis Rate (FSR) with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: during HDBR period
  Measurement of protein turnover.
Changes in sleep quality with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Sleep quality will be assessed using a 3-electrode electroencephalogram (EEG) Sleep Profiler and a wrist worn actigraphy.
Changes in sleep architecture with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Using 3-electrode electroencephalogram (EEG) Sleep Profiler electrical patterns of brain activity will be measured in order to assess sleep cycles and sleep stages.
Changes in frailty status with HDBR with and without exercise countermeasure. | Throughput the 26-day study period: at Baseline, HDBR and Recovery periods
  CLSA-FI questionnaire
Changes in the gut microbiome with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  To assess gut microbiome, stool samples will be collected and targeted sequencing of the variable regions 4 and 5 (V4-V5) of the 16S ribosomal RNA gene will be performed on an Illumina MiSeq.
Changes in the constitution of the oral microbiome with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  To assess oral microbiome, saliva samples will be collected and targeted sequencing of the variable regions 4 and 5 (V4-V5) of the 16S ribosomal RNA gene will be performed on an Illumina MiSeq.
Changes in physical performance with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Short Physical Performance Battery test
Changes in physical performance with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Timed-up-and-Go test
Changes in dynamic balance with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Four-square step test
Changes in bone markers with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  The following bone markers will be assessed using ELISA kits:
  * Total osteocalcin
  * Undercarboxylated osteocalcin
  * Sclerostin
  * NTX (N-terminal Telopeptide)
  * CTX (C-terminal telopeptide)
  * Bone Specific Alkaline Phosphatase (BSAP)
  * Procollagen type 1 amino-terminal propeptide (P1NP)
Changes in growth factors with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  The following growth factors will be measured with Multiplex:
  * Basic fibroblast growth factor
  * Granulocyte colony-stimulating factor (G-CSF)
  * Granulocyte-macrophage colony-stimulating factor (GM-CSF)
  * Platelet-derived growth factor BB (PDGF-BB)
  * Transforming growth factor β (TGF-β)
  * Vascular endothelial growth factor (VEGF)
Changes in cytokines with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  The following cytokines will be measured with Multiplex:
  * Eotaxin
  * Interferon gamma (IFN-γ)
  * IL-1β, IL-1Ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17
  * Tumour necrosis factor (TNF-α)
  * Interferon gamma- induced protein 10 (IP-10)
  * Monocyte chemoattractant protein 1 (MCP-1)
  * Macrophage inflammatory protein-1α (MIP-1α)
  * Macrophage inflammatory protein-1β (MIP-1β)

SECONDARY OUTCOMES:
Changes in neuromotor function with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Neuromuscular activity will be assessed using electromyography.
Changes in aerobic capacity with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Bicycle Ergometer Test
Changes in body composition with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline and Recovery periods
  Lean muscle and fat mass will be assess using dual energy X-ray absorptiometry.
Changes in insulin sensitivity with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  Will measure excursion curves of glucose and insulin.
Changes in neuronal factors with HDBR with and without exercise countermeasure. | Throughout the 26-day study period: at Baseline, HDBR and Recovery periods
  The following bone markers will be assessed using ELISA kits:
  * Neurofilament light chain
  * Glial fibrillary acidic protein
  * Myelin basic protein
  * Total tau
  * Aβ1-40
  * Aβ1-42
  * BDNF

CONTACTS AND LOCATIONS:
Overall Officials: José A. Morais, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University
Locations (1):
- Royal Victoria Hospital - Glen site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mastrandrea CJ, Hajj-Boutros G, Sonjak V, Hedge ET, Gouspillou G, Hughson RL, Morais JA. Exercise attenuates bed rest-induced increases in insulin resistance while alpha-klotho increases in 55 to 65 year-old women and men. Sci Rep. 2025 Jul 24;15(1):26927. doi: 10.1038/s41598-025-12770-5. PMID 40707556
- [Derived] Balbim GM, Falck RS, Barha CK, Tai D, Best JR, Hajj-Boutros G, Madden K, Liu-Ambrose T. Exercise counters the negative impact of bed rest on executive functions in middle-aged and older adults: A proof-of-concept randomized controlled trial. Maturitas. 2023 Oct 17;179:107869. doi: 10.1016/j.maturitas.2023.107869. Online ahead of print. PMID 39491057
- [Derived] Blaber AP, Sadeghian F, Naz Divsalar D, Scarisbrick IA. Elevated biomarkers of neural injury in older adults following head-down bed rest: links to cardio-postural deconditioning with spaceflight and aging. Front Hum Neurosci. 2023 Sep 26;17:1208273. doi: 10.3389/fnhum.2023.1208273. eCollection 2023. PMID 37822710